CLINICAL TRIAL: NCT07317648
Title: ClearSight NextGen System Clinical Development Study
Brief Title: ClearSight NextGen1 Study
Status: Recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-01
Record Dates: First submitted 2025-11-21; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adult OR patients with planned or existing arterial blood pressure monitoring
  Interventions: Device: ClearSight NextGen system

INTERVENTIONS:
Device: ClearSight NextGen system — Study devices will be applied to subjects for monitoring for the duration of the procedure.

SUMMARY:
A prospective, non-randomized single arm study using the investigational ClearSight NextGen (CSNG) system in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age ≥ 18 years
3. Planned or existing monitoring with an arterial catheter as part of standard of care
4. Patient scheduled to undergo surgery with general anesthesia lasting > 2 hours

Exclusion Criteria:

1. Any significant disfigurement or prior injury to a participant's finger that is intended to be used for monitoring with the study finger cuffs
2. Known left-right difference in blood pressure
3. Extreme contraction of the smooth muscles in the arteries and arterioles of the lower arm and hand, such as may be present in patients with Raynaud's disease
4. Patients deemed not suitable for the study at the discretion of the Investigator
5. Participation in another study that clinically interferes with the current study
6. Treatment with an intra-aortic balloon pump
7. Pregnancy
8. Cardiac surgery including bypass period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ≥ 18 years scheduled to undergo surgery with general anesthesia lasting >2 hours; with planned or existing monitoring with an arterial catheter as part of standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Data Collection for Development of ClearSight NextGen System | Monitoring during surgery, for up to approximately 4 hours.
  The objective of the study is to collect blood pressure data using the investigational CSNG system alongside CE-Marked ClearSight and FloTrac devices in adult subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- York Teaching Hospitals NHS Foundation Trust, York, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No